CLINICAL TRIAL: NCT00929318
Title: Clinical Investigations on Cytokin-Gradients in Hypo/Euthyroid Patients. Evaluation of Expression of Different Pro-and Anti-Inflammatory Cyto-/Chemokines in Skin Wounds After Surgery of Benign Goitres (Struma Multinodosa) or Malignant Diseases of Thyroid Gland (Papillary Thyroid Carcinoma) in Correlation to the Status of Wound Healing of the Neck Wound
Brief Title: Influence of Thyroid Hormones on the Woundhealing Process
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Prof. Dr Georg FW Scheumann, Medizinische Hochschule Hannover
Allocation: Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: MHH-THY-WH-09
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2009-06

CONDITIONS: Thyroid Neoplasms; Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- benign (Active Comparator): patients after surgery because of a benign disease
  Interventions: Procedure: blood sampling
- DTC (Active Comparator): Patients after thyroidectomy because of papillary carcinoma of the thyroid gland
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling
Procedure: blood sampling
  Arms: benign

SUMMARY:
Main goal of this clinical investigation is to investigate different cytokines in wound fluids of euthyroid vs. hypothyroid patients. As a primary endpoint we want to evaluate if different cytokine levels in euthyroid vs. hypothyroid patients exist and to what extent these cytokines differ. Our targeted cytokines are: IL6, IL10, TNFa and MCP-1. From the literature these 4 factors seem to be the most reasonable to measure and to focus on. Additionally we focus on these 4 factors for financial reasons, technically there wouldn't be a problem to measure more, which is correlated with higher costs. Besides, more than 6 factors would mean larger amounts of sample fluids needed, which would cause technical problems. These factors don't have to change in the same direction. Secondarily, we believe that differences in cytokine profiles of hypothyroidism vs. euthyroidism will correlate to differences in duration and clinical characteristics of the wound healing process.

ELIGIBILITY:
Inclusion Criteria:

* Near total or total thyroidectomy because of struma multinodsa (nodular goiter) with or without substitution of thyroid hormone after operation
* Total thyroidectomy because of papillary carcinoma of thyroid gland (T1/T2 carcinoma, N1, M0) with planned radio-ablative therapy (RAT) without or with rhTSH

Exclusion Criteria:

* Pat< 18 years
* Immune disease of thyroid gland (Graves disease)
* Severe immunodeficiency
* Immunosuppressive medication because of solid Organ transplantation
* Hepatitis A/B/C or HIV
* All exclusion criteria for any surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Evidence for different cytokine levels in euthyroid vs hypothyroid condition confirmed by bood serum samples | 21 days after surgery

SECONDARY OUTCOMES:
Differences in duration and clinical characteristics of the wound healing process verified by a modified ASEPSIS score. | 21 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hoochschule Hannover, Allgemein-, Viszeral-und Transplantationscirurgie OE 6220, Hanover, Germany